CLINICAL TRIAL: NCT00485875
Title: An Open-Label, Multicenter, Pilot Study of the Safety and Efficacy of Transitioning From a Stimulant Medication to Atomoxetine in Pediatric and Adolescent Outpatients With DSM-IV Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy of Switching From a Stimulant Medication to Atomoxetine in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7953; B4Z-MC-LYCI
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride

SUMMARY:
The purpose of this study is to assess changes in ADHD symptoms and tolerability of medication in children and adolescents switching from a stimulant to atomoxetine.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 6 years of age and not yet be 18 years of age at the completion of visit 6
* Patients must meet DSM-IV diagnostic criteria for ADHD (any subtype)
* Patients must have laboratory results showing no significant abnormalities (significant would include laboratory deviations requiring acute medical intervention or further medical evaluation)
* Patients must be of normal intelligence as assessed by the investigator (that is, without a general impairment of intelligence and likely, in the investigator's judgment, to achieve a score of greater than or equal to 70 on a IQ test)
* Patients must be able to swallow capsules

Exclusion Criteria:

* Patients who weigh less than 22 kg or more than 70 kg at study entry
* Patients who have a history of Bipolar I or Bipolar II Disorder, psychosis, or a pervasive developmental disorder
* Patients with a history of any seizure disorder (other than febrile seizures) or prior EEG abnormalities related to epilepsy, or patients who have taken (or are currently taking) anticonvulsants for seizure control
* Patients with a history of severe allergies to more than one class of medication, or multiple adverse drug reactions
* Patients who have glaucoma

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2004-06; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Assess the change in ADHD symptoms when switching from stimulant medication to atomoxetine among patients who cannot tolerate or do not respond to stimulants and require a medication change

SECONDARY OUTCOMES:
Assess whether there are statistically significant differences in ADHD symptom measures after a patient changes from a stimulant medication to atomoxetine
Assess the safety and tolerability of atomoxetine alone compared with stimulant medications alone and during the time of switch (stimulant plus atomoxetine) as assessed by AEs elicited during open-ended questioning.
Compare atomoxetine and stimulant medications on other secondary measures, including parent preference
Assess whether there is a significant change in problem behaviors related to ADHD after switching from stimulant medication to atomoxetine
Assess the change in inattentive and hyperactive symptoms among these same patients

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-582-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com